CLINICAL TRIAL: NCT00830804
Title: A Pilot Efficacy and Safety Trial of Raltegravir Plus Darunavir/Ritonavir for Treatment-Naive HIV-1-Infected Subjects
Brief Title: Safety and Effectiveness of Raltegravir Plus Darunavir/Ritonavir in Treatment-Naive HIV-Infected Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5262; 1U01AI068636 (NIH)
Record Dates: First submitted 2009-01-26; First posted 2009-01-28 (Estimated); Results first posted 2011-10-10 (Estimated); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: HIV-1 Infections
Keywords: Treatment Naive
MeSH Terms: interventions — Raltegravir Potassium; Darunavir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RAL + DRV/RTV (Experimental): Raltegravir (400 mg BID) plus Darunavir/Ritonavir (800 mg/100 mg QD) for 52 weeks
  Interventions: Drug: Raltegravir; Drug: Darunavir/Ritonavir

INTERVENTIONS:
Drug: Raltegravir — 400 mg tablet taken orally twice daily
  Other Names: RAL
Drug: Darunavir/Ritonavir — 800 mg Darunavir/100 mg Ritonavir tablet taken orally once daily
  Other Names: DRV/RTV

SUMMARY:
The purpose of this study is to assess the effectiveness and safety of an antiretroviral therapy (ART) regimen consisting of raltegravir (RAL) and darunavir (DRV)/ritonavir (RTV) as first-line therapy in treatment-naïve participants.

DETAILED DESCRIPTION:
Despite the remarkable strides made in the treatment of HIV-1-infected persons over the last decade, current first-line ART regimens are imperfect. The ideal combination, unlike some current first-line options, would have uncompromised efficacy in the presence of transmitted drug-resistant variants. The primary purpose of this study is to estimate the cumulative proportion of ART-naive participants experiencing virologic failure at or prior to week 24 after initiating raltegravir (RAL) plus darunavir/ritonavir (DRV/RTV).

The study will last 52 weeks. All participants will follow the same treatment schedule and take RAL plus DRV/RTV orally daily for the duration of the trial.

After entry, all participants will have scheduled visits at weeks 1, 4, 12, 24, 36, 48, and 52. Medical/medication history, blood and urine collection, and liver function tests will occur at screening. A targeted physical exam and concomitant medications history will occur at all study visits. Blood and urine collection and liver function tests will occur at most study visits. For females, a pregnancy test will occur at screening and study entry.

RAL and DRV were provided by the study. RTV was not provided by the study.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1-infected
* Plasma HIV-1 RNA of at least 5,000 copies/mL within 90 days prior to study entry
* HIV genotype (for reverse transcriptase and protease) performed at any time prior to study entry. More information on this criterion can be found in the protocol.
* ARV drug-naive. More information on this criterion can be found in the protocol.
* Negative result from a hepatitis B surface antigen test performed within 90 days prior to study entry
* Agree to use one form of medically-accepted contraceptive throughout the study and for 60 days after stopping study treatment. More information on this criterion can be found in the protocol.

Exclusion Criteria:

* Serious illness requiring systemic treatment and/or hospitalization for at least 7 days prior to study. More information on this criterion can be found in the protocol.
* Screening HIV genotype obtained any time prior to study entry with more than one DRV resistance-associated mutation [RAM] (V11I, V32I, L33F, I47V, I50V, I54L, I54M, T74P, I84V, and L89V) or L76V alone
* Known major integrase inhibitor RAM(s), including N155H, Q148H/R/K, Y143C/R, and G140S
* Severe renal insufficiency requiring hemodialysis or peritoneal dialysis
* Treatment with immunomodulators within 30 days prior to study entry. More information on this criterion can be found in the protocol.
* Current medications that are prohibited with any study medications. More information on this criterion can be found in the protocol.
* Known allergy/sensitivity to study drugs or their formulations. A history of sulfa allergy is not an exclusion.
* Active drug or alcohol use or dependence that, in the opinion of the investigator, would interfere with the study.
* Certain abnormal laboratory results. More information on this criterion can be found in the protocol.
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2009-04; Primary Completion 2010-02 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J. Eron, Jr., MD, Study Chair — University of North Carolina, Chapel Hill
Locations (22):
- United States (22):
  - AlabamaTherapeutics CRS, Birmingham, Alabama
  - Stanford CRS, Palo Alto, California
  - Ucsd, Avrc Crs, San Diego, California
  - Ucsf Aids Crs, San Francisco, California
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Georgetown University CRS, Washington D.C., District of Columbia
  - Northwestern University CRS, Chicago, Illinois
  - Beth Israel Deaconess Med Center, Boston, Massachusetts
  - Brigham and Women's Hosp. ACTG CRS, Boston, Massachusetts
  - Washington U CRS, St Louis, Missouri
  - AIDS Community Health Ctr. ACTG CRS, Rochester, New York
  - Unc Aids Crs, Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS, Durham, North Carolina
  - Univ. of Cincinnati CRS, Cincinnati, Ohio
  - Case CRS, Cleveland, Ohio
  - MetroHealth CRS, Cleveland, Ohio
  - The Ohio State Univ. AIDS CRS, Columbus, Ohio
  - Hosp. of the Univ. of Pennsylvania CRS, Philadelphia, Pennsylvania
  - University of Pittsburgh CTU, Pittsburgh, Pennsylvania
  - The Miriam Hospital, Providence, Rhode Island
  - Vanderbilt Therapeutics CRS, Nashville, Tennessee
  - Houston AIDS Research Team, Houston, Texas

REFERENCES:
- [Background] Capetti AF, Piconi S, Landonio S, Rizzardini G, Perno CF. Is dual therapy with raltegravir and protease inhibitors a feasible option in rescue strategy in HIV-1 infection? J Acquir Immune Defic Syndr. 2009 Feb 1;50(2):233-4. doi: 10.1097/QAI.0b013e31818c7e8e. No abstract available. PMID 19155770
- [Background] Long MC, King JR, Acosta EP. Pharmacologic aspects of new antiretroviral drugs. Curr HIV/AIDS Rep. 2009 Feb;6(1):43-50. doi: 10.1007/s11904-009-0007-y. PMID 19149996
- [Background] Vermeir M, Lachau-Durand S, Mannens G, Cuyckens F, van Hoof B, Raoof A. Absorption, metabolism, and excretion of darunavir, a new protease inhibitor, administered alone and with low-dose ritonavir in healthy subjects. Drug Metab Dispos. 2009 Apr;37(4):809-20. doi: 10.1124/dmd.108.024109. Epub 2009 Jan 8. PMID 19131522
- [Derived] Taiwo B, Zheng L, Gallien S, Matining RM, Kuritzkes DR, Wilson CC, Berzins BI, Acosta EP, Bastow B, Kim PS, Eron JJ Jr; ACTG A5262 Team. Efficacy of a nucleoside-sparing regimen of darunavir/ritonavir plus raltegravir in treatment-naive HIV-1-infected patients (ACTG A5262). AIDS. 2011 Nov 13;25(17):2113-22. doi: 10.1097/QAD.0b013e32834bbaa9. PMID 21857490

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited from 22 U.S. sites from April 2009 to August 2009.
Pre-assignment Details: Study participants were HIV-1-infected, antiretroviral(ARV)-naive men and women, 18 years and older with plasma HIV-1 RNA >= 5000 copies/ml. One enrolled participant never started study treatment.
Period: Overall Study
Arm/Group | RAL + DRV/RTV
Started | 112 (113 subjects enrolled. One subject never started study treatment and was excluded in all analysis.)
Completed | 97
Not Completed | 15
Not completed — Lost to Follow-up | 4
Not completed — Death | 1
Not completed — Unable to get to clinic | 7
Not completed — Consent withdrawn | 2
Not completed — Unwilling to adhere to study requirement | 1

BASELINE CHARACTERISTICS:
Groups:
- RAL+DRV/RTV: Raltegravir (400 mg BID) plus Darunavir/Ritonavir (800 mg/100 mg QD) for 52 weeks
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 112
Age, Continuous [Median (Full Range); unit: years] — Age (in years) of participants at study entry
  years | 36 (11) [19 to 66]
Age, Customized [Number; unit: participants] — Age (in years) of participants at study entry
  participants
    18-29 | 33
    30-39 | 38
    40-49 | 25
    50-59 | 12
    60-69 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 112

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Virologic Failure After Initiating RAL Plus DRV/RTV at or Prior to Week 24
Description: Virologic failure is defined as: at week 12, confirmed plasma HIV-1 RNA >= 1000 copies/ml or confirmed rebound from the week 4 value by >0.5 log10 copies/ml (for subjects with week 4 value <= 50 copies/ml, confirmed rebound to >50 copies/ml); at week 24 or later, confirmed value > 50 copies/ml. Viral load confirmation was scheduled 7-35 days after initial virologic failure. The proportion was estimated using Kaplan-Meier method. An adaptation of Greenwood's variance estimate was used in constructing the confidence interval.
Time Frame: From start of study treatment to week 24
Population: All participants who started study treatment were included. The intent-to-treat approach was used, ignoring whether a participant was on or off treatment at the time of HIV-1 RNA measurement and censoring follow-up if a participant was lost-to-follow-up without previously meeting the definition of virologic failure.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 112
Proportion of participants | 0.16 [0.10 to 0.24]

2. Secondary Outcome: Proportion of Participants With Virologic Failure or Off Study Treatment Regimen or Death at or Prior to Week 24
Description: The proportion of participants with virologic failure (see primary outcome measure for definition) and/or premature treatment discontinuation/modification and/or death was estimated using Kaplan-Meier method. An adaptation of Greenwood's variance estimate was used in constructing the confidence interval.
Time Frame: From start of study treatment to Week 24
Population: All participants who started study treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 112
Proportion of participants | 0.21 [0.14 to 0.29]

3. Secondary Outcome: Change in Plasma HIV-1 RNA From Baseline to Week 1
Description: Results report the week 1 change from baseline (week 1 - baseline) in HIV-1 RNA. Baseline HIV-1 RNA was computed as the mean of the log10 HIV-1 RNA values at pre-entry and study entry.
Time Frame: Baseline and week 1
Population: Analyis was based on an intent-to-treat approach, ignoring whether a participant was on or off study treatment at the time the sample for HIV-1 RNA was obtained.
Measure: Median (Inter-Quartile Range); unit: log10 copies/ml
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 112
log10 copies/ml | -1.67 [-1.93 to -1.42]

4. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA < 50 Copies/ml or <200 Copies/ml at Week 24
Description: Results report the percentage of participants with plasma HIV-1 RNA < 50 copies/ml or <200 copies/ml at week 24.
Time Frame: From start of study treatment to week 24
Population: All participants who started study treatment were included. An intent-to-treat approach was used ignoring participants who were off-study or with missing HIV-1 RNA at week 24.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 107
proportion of participants
  With HIV-1 RNA < 50 copies/ml | 0.79 [0.70 to 0.86]
  With HIV-1 RNA < 200 copies/ml | 0.93 [0.87 to 0.97]

5. Secondary Outcome: Proportion of Participants With Plasma HIV-1 RNA <50 Copies/ml or <200 Copies/ml at Week 48
Description: Results report the percentage of participants with plasma HIV-1 RNA <50 copies/ml or <200 copies/ml at week 48.
Time Frame: From start of study treatment to week 48
Population: All participants who started study treatment were included. An intent-to-treat approach was used ignoring participants who were off study treatment or with missing HIV-1 RNA at week 48.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 100
proportion of participants
  With HIV-1 RNA < 50 copies/ml | 0.71 [0.61 to 0.79]
  With HIV-1 RNA < 200 copies/ml | 0.86 [0.78 to 0.92]

6. Secondary Outcome: Proportion of Participants Who Experienced Signs/Symptoms or Laboratory Toxicities Grade 3 or Higher, or of Any Grade Which Led to a Permanent Change or Discontinuation of Study Treatment
Description: Signs, symptoms and laboratory values were graded according to the Division of AIDS Adverse Event Grading System. Results report the percentage of participants who had grade 3 or higher events, or events of any grade which led to a permanent change or discontinuation of study treatment, which occurred any time from start of treatment to end of treatment.
Time Frame: From start of study treatment to week 52
Population: All participants who started study treatment were included in the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 112
proportion of participants | 0.20 [0.13 to 0.28]

7. Secondary Outcome: Number of Participants With Pretreatment Drug Resistance
Description: Results report the number of participants who had resistance to non-nucleoside reverse transciptase inhibitors (NNRTI), nucleoside reverse transciptase inhibitors (NRTI) and protease inbitors (PI) based on genotypic resistance testing done prior to participant's entry into the study. Participants are classified into one (and only one category) based on the maximum number of drug class resistance seen for the participant.
Time Frame: At screening
Population: All participants who started study treatment were included in the analysis.
Measure: Number; unit: participants
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 112
participants
  With NNRTI mutations only | 9
  With NRTI mutations only | 8
  With Both NNRTI and NRTI mutations | 1
  With PI mutations only | 2
  With PI, NNRTI and NRTI mutations | 1
  No Resistance Detected | 91

8. Secondary Outcome: Number of Participants With Integrase Drug Resistance at Virologic Failure
Description: Results report the number of participants who had integrase resistance mutation(s) detected at the time of virologic failure.
Time Frame: From 12 weeks after starting study treatment to week 52
Population: Only those participants who had virologic failure (see primary outcome measure for definition) and who had successful integrase genotyping at failure were included in the analysis.
Measure: Number; unit: participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 25
participants | 5

9. Secondary Outcome: Number of Participants With Protease Drug Resistance at Virologic Failure
Description: Results report the number of participants who had protease resistance mutation(s) detected at the time of virologic failure.
Time Frame: From 12 weeks after starting study treatment to week 52
Population: Only those participants who had virologic failure (see primary outcome measure for definition) and who had successful protease genotyping at failure were included in the analysis.
Measure: Number; unit: participants
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 23
participants | 0

10. Secondary Outcome: Number of Participants With Perfect Overall Adherence by Self Report
Description: At each study visit, adherence was measured in terms of the number of missed doses each participant had over a 4-day recall for each drug. Adherence for all study visit weeks were combined for an overall measure of adherence. Participants who had zero missed doses on all weeks in all drugs while on study were classified as having an overall "perfect" adherence.
Time Frame: From one week after starting study treatment to week 52
Population: All participants who started study treatment were included in the analysis.
Measure: Number; unit: participants
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 112
participants | 95

11. Secondary Outcome: Changes in Fasting Total Cholesterol, High-density Lipoprotein and Triglyceride at Week 24
Description: Results report the week 24 change from week 0 (week 24 - week 0) fasting total cholesterol, high-density lipoprotein and triglyceride.
Time Frame: From start of study treatment through week 24
Population: Only those participants who started study treatment and who had fasting lipid measurements at week 24 and week 0 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 94
mg/dL
  Fasting Total Cholesterol | 31.5 [12 to 46]
  Fasting High-density Lipoprotein | 6.5 [1 to 15]
  Fasting Triglyceride | 24.5 [-6 to 64]

12. Secondary Outcome: Change in Fasting Low-density Lipoprotein at Week 24
Description: Results report the week 24 change from week 0 (week 24 - week 0) fasting low-density lipoprotein (LDL). For participants whose calculated fasting LDL and direct fasting LDL were both reported, only the calculated fasting LDL was used. Direct fasting LDL was reported when the participant had high fasting triglyceride.
Time Frame: From start of study treatment through week 24
Population: as for outcome 11
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 82
mg/dL | 16.0 [5 to 36]

13. Secondary Outcome: Changes in Fasting Total Cholesterol, High-density Lipoprotein and Triglyceride at Week 48
Description: Results report the week 48 change from week 0 (week 48 - week 0) fasting total cholesterol, high-density lipoprotein and triglyceride.
Time Frame: From start of study treatment through week 48
Population: Only those participants who started study treatment and who had fasting lipid measurements at week 48 and week 0 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 85
mg/dL
  Fasting Total Cholesterol | 30 [10 to 59]
  Fasting High-density Lipoprotein | 9 [2 to 17]
  Fasting Triglyceride | 23 [-31 to 81]

14. Secondary Outcome: Change in Fasting Low-density Lipoprotein at Week 48
Description: Results report the week 48 change from week 0 (week 48 - week 0) fasting low-density lipoprotein (LDL). For participants whose calculated fasting LDL and direct fasting LDL were both reported, only the calculated fasting LDL was used. Direct fasting LDL was reported when the participant had high fasting triglyceride.
Time Frame: From start of study treatment through week 48
Population: as for outcome 13
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 70
mg/dL | 17 [2 to 33]

15. Secondary Outcome: Change in CD4 Count at Week 48
Description: Results report the week 48 change from baseline (week 48 - baseline) in CD4 count. Baseline CD4 count was computed as the mean of CD4 count values at pre-entry and study entry.
Time Frame: From start of study treatment through week 48
Population: Only those participants who started study treatment and who have values at baseline and at week 48 were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: cells/mm3
Arm/Group | RAL + DRV/RTV
Number analyzed (Participants) | 100
cells/mm3 | 200 [114 to 318]

16. Secondary Outcome: Plasma Trough Concentration of Raltegravir
Description: Plasma trough concentrations (ng/ml) of Raltegravir (RAL) below the detection limit (10 ng/ml) were replaced by half the corresponding lower limit of quantitation. Geometric mean of trough concentrations obtained within the prescribed trough time (within 9-15 hours after the last RAL dose) was computed for each participant. For participants who experienced virologic failure (see primary outcome measure definition), only those concentrations on or before virologic failure confirmation were used in the geometric mean computation.
Time Frame: From start of study treatment to week 52
Population: Participants who started study treatment and who have at least one RAL plasma trough concentration obtained within 9-15 hours after the last RAL dose were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 103
ng/ml | 117 [52 to 250]

17. Secondary Outcome: Plasma Trough Concentration of Darunavir
Description: Plasma trough concentrations (ng/ml) of Darunavir (DRV) below the detection limit (50 ng/ml) were replaced by half the corresponding lower limit of quantitation. Geometric mean of trough concentrations obtained within the prescribed trough time (within 20-28 hours after the last DRV dose) was computed for each participant. For participants who experienced virologic failure (see primary outcome measure definition), only those concentrations on or before virologic failure confirmation were used in the geometric mean computation.
Time Frame: From start of study treatment to week 52
Population: Participants who started study treatment and who have at least one DRV plasma trough concentration obtained within 20-28 hours after the last DRV dose were included in the analysis.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | RAL+DRV/RTV
Number analyzed (Participants) | 83
ng/ml | 1218 [789 to 1809]

ADVERSE EVENTS:
Time Frame: From start of study treatment to week 52
Description: Expedited adverse event (AE) reporting followed Intensive Division of AIDS (DAIDS) Reporting Level, which included AEs resulting in death, congenital anomalies, fetal losses, significant disabilities, requiring hospitalization, and >=grade 3 AEs defined by the "DAIDS Table for Grading the Severity of Adult and Pediatric AEs", V1.0, 12/2004.
Arm/Group | RAL+DRV/RTV
Serious Adverse Events (participants affected / at risk) | 13/112
Other Adverse Events (participants affected / at risk) | 78/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RAL+DRV/RTV (N=112)
Diarrhoea (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Injection site reaction (General disorders) | 1
Bronchitis (Infections and infestations) | 1
Perirectal abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Alcohol poisoning (Injury, poisoning and procedural complications) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Convulsion (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Substance abuse (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | RAL+DRV/RTV (N=112)
Nausea (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 11
Aspartate aminotransferase increased (Investigations) | 15
Blood cholesterol (Investigations) | 45
Blood glucose abnormal (Investigations) | 8
Blood sodium decreased (Investigations) | 6
Blood uric acid increased (Investigations) | 9
Low density lipoprotein abnormal (Investigations) | 34
Neutrophil count decreased (Investigations) | 14
White blood cell count decreased (Investigations) | 8
Depression (Psychiatric disorders) | 7

LIMITATIONS AND CAVEATS:
This is a single-arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trial Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.